CLINICAL TRIAL: NCT01823185
Title: Bedside Testing of the CYP2C19 Gene to Asses Effectiveness of Clopidogrel in Coronary Artery Disease Patients Treated With Percutaneous Coronary Intervention : Individualized Antiplatelet Drugs Treatment to Improve Prognosis
Brief Title: Bedside Testing of CYP2C19 Gene for Treatment of Patients With PCI With Antiplatelet Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Collaborators: King Fahad Armed Forces Hospital (Other Government); Dammam Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STGUD005
Record Dates: First submitted 2013-03-19; First posted 2013-04-04 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Coronary Artery Disease; Myocardial Infarction; Heart Disease; Vascular Disease; Angina Pectoris; Cardiovascular Disease; Ischemia; Infarction; Embolism; Thrombosis; Chest Pain
Keywords: Clopidogrel; Ticagrelor; Prasugrel; Platelet aggregation inhibitor; Dammam University; King Fahd Hospital; Purinergic P2 receptor Antagonists
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction; Heart Diseases; Vascular Diseases; Angina Pectoris; Cardiovascular Diseases; Ischemia; Infarction; Embolism; Thrombosis; Chest Pain | interventions — Clopidogrel; Ticagrelor; Prasugrel Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clopidogrel (Active Comparator): CYP2C19 genotyping will be carried out at the end of the study period. Clopidogrel will be used for treatment for one year according to local protocol. Patients will receive clopidogrel 75 mg per day.
  Interventions: Drug: clopidogrel
- Ticagrelor or prasugrel (Experimental): Ticagrelor (90 mg twice daily) or prasugrel ( 10mg once daily or 5mg once daily if the patient older than 75 years or a body weight < 60kg) according to local protocol.
  Interventions: Drug: Ticagrelor or prasugrel

INTERVENTIONS:
Drug: clopidogrel — Genotyping will be carried out using Spartan genotyping System on all intervention group and those patients who do not carry the CYP2C19 allele 2 or 3 will be given clopidogrel (75 mg per day) while all patients who carry the CYP2C19 allele 2 or 3 will be prescribed Ticagrelor (90 mg twice daily) or prasugrel ( 10mg once daily or 5mg once daily if the patient older than 75 years or a body weight < 60kg) according to local protocol.
  Other Names: Clavix
  Arms: Clopidogrel
Drug: Ticagrelor or prasugrel — ticagrelor (90 mg twice daily) or prasugrel ( 10mg once daily or 5mg once daily if the patient older than 75 years or a body weight < 60kg) according to local protocol.
  Other Names: Brilinta; Prasuvas
  Arms: Ticagrelor or prasugrel

SUMMARY:
Clopidogrel is crucial as antiplatelet treatment in patients undergoing percutaneous coronary intervention (PCI) with stent implantation and during one year after PCI, to prevent atherothrombotic complications. However, clopidogrel is ineffective in certain patients due to genetic mutation in CYP2C19 gene a specific enzyme in the liver required for metabolism of clopidogrel. Therefore, the purpose of this study is to test these patients genetically at bedside and prescribe an alternative drug such as Ticagrelor (90 mg twice daily) or prasugrel ( 10mg once daily or 5mg once daily if the patient older than 75 years or a body weight < 60kg) if they are carriers of the allele 2 or 3 of the mutated gene.

DETAILED DESCRIPTION:
Clopidogrel is crucial as antiplatelet treatment in patients undergoing percutaneous coronary intervention (PCI) with stent implantation and during one year after PCI, to prevent atherothrombotic complications. Clopidogrel is converted into its active metabolite by Cytochrome P2C19 (CYP2C19). However 30 % of the Saudi population is carrier of the non functional CYP2C19*2 or *3 alleles having an impaired CYP2C19 capacity, resulting in decreased effectiveness of Clopidogrel. These patients have a 42% higher risk for major cardiovascular events (MACE) compared to non carriers. Further 50 % of the MACE occurs in the first 48 hours. Therefore Ticagrelor (90 mg twice daily) or prasugrel ( 10mg once daily or 5mg once daily if the patient older than 75 years or a body weight < 60kg) whose actions are not dependent on conversion by CYP2C19 may be an alternative only in carriers of the non functional CYP2C19*2 or *3 alleles. This might be cost effective and prevent patients form MACE. Therefore the objective of this study is to assess the efficacy, complication free survival, safety and cost-effectiveness of the CYP2C19 genotype guided antiplatelet treatment strategy, using clopidogrel or prasugrel (or Ticlid). All participants will be followed for one year using follow up questionnaires.

ELIGIBILITY:
Male & female age 18-70 years

Inclusion Criteria:

* Patient presents with acute myocardial infarction of more than 30 minutes and less than 12 hours
* Patient eligible for PCI

Exclusion Criteria:

* Life expectancy of less than one year
* Previously Known genotype
* Receiving chemotherapy for malignancy
* On dialysis or receiving immunosuppressive therapy or have autoimmune disease
* Hepatic impairment
* History of bleeding diathesis
* Receiving vitamin K antagonist therapy
* Confirmed hypertension
* Out of normal range platelet count
* History of major surgery
* Severe trauma or fracture
* Pregnancy and lactation
* Concomitant use of simvastatin, cytochrome P450 3A4 inhibitors or inducers
* Hypersensitivity to clopidogrel or ticagrelor or prasugrel

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2013-03; Primary Completion 2016-01 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
cardiovascular event | 1 year
  The primary end point is the number of patients who develop adverse major cardiovascular event which include recurrent myocardial infarction, non-fatal stroke, cardiovascular mortality, severe ischemia, major bleeding at 30days after PCI.

SECONDARY OUTCOMES:
Mortality | 30 days and 1 year
  Secondary efficacy endpoints are the number of patients who either died , died from cardiovascular death, from cerebrovascular death, developed recurrent MI, stent thrombosis, underwent urgent target vessel revascularization, developed stroke or combination of above

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah M Al-Rubaish, MD, Principal Investigator — Imam Abdulrahman Bin Faisal University; Amein K Al-Ali, PhD, Study Director — Imam Abdulrahman Bin Faisal University
Locations (4):
- Saudi Arabia (4):
  - Prince Sultan Cardiac center, Al-Hasa
  - Saud Al-Babtain Cardiac Center, Dammam
  - King Fahd Military Medical Complex, Dammam
  - King Fahd University Hospital, Khobar

REFERENCES:
- [Derived] Al-Rubaish AM, Al-Muhanna FA, Alshehri AM, Al-Mansori MA, Alali RA, Khalil RM, Al Faraidy KA, Cyrus C, Sulieman MM, Vatte C, Claassens DMF, Ten Berg JM, Asselbergs FW, Al-Ali AK. Bedside testing of CYP2C19 gene for treatment of patients with PCI with antiplatelet therapy. BMC Cardiovasc Disord. 2020 Jun 3;20(1):268. doi: 10.1186/s12872-020-01558-2. PMID 32493215